CLINICAL TRIAL: NCT01526720
Title: The Verona Newly Diagnosed Type 2 Diabetes Study. Construction of a Biobank of Diabetes Related Genotypes and Phenotypes
Brief Title: The Verona Newly Diagnosed Type 2 Diabetes Study
Acronym: VNDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: European Foundation for the Study of Diabetes (Other); Ministry of Education, Universities and Research, Italy (Other)
Responsible Party: Principal Investigator, Riccardo Bonadonna, Professor, Universita di Verona
Other Study IDs: CE-955
Record Dates: First submitted 2012-01-27; First posted 2012-02-06 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Beta cell function; Insulin sensitivity; Genetics of diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood Serum Plasma Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: Diabetic: Newly diagnosed type 2 diabetic patients (i.e. diagnosis made no more than 6 months before recruitment)
- Group B: Relatives: Relatives of patients with potentially monogenic newly diagnosed type 2 diabetes

SUMMARY:
Type 2 diabetes mellitus is a complex disease whose clinical phenotype results from the variable combination of genetic and nongenetic factors. The aim of the present study is to investigate the network linking phenotypes and genotypes in patients with newly diagnosed type 2 diabetes mellitus. In selected cases, in which clinical evidence hints at possible monogenic basis of the disease, the genotype and the phenotype of relatives also will be assessed to elucidate further the etiology of the disease.

DETAILED DESCRIPTION:
The Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) is an ongoing study aiming at building a biobank of patients with newly diagnosed type 2 diabetes mellitus. All patients referred to the Division of Endocrinology and Metabolic Diseases of University of Verona School of Medicine, whose diabetes has been diagnosed in the last six months, are asked to participate in this research. The clinical evidence on which the diagnosis of type 2 diabetes has been made is reviewed and the diagnosis confirmed, according to the current criteria of American Diabetes Association. Patients already treated with antidiabetic drugs undergo a treatment washout of at least one week before metabolic tests are performed. Among the exclusion criteria are age > 75 years, non-Italian ancestry, insulin treatment, presence of anti-GAD antibodies, malignancies, and any condition severely impairing liver and/or kidney function.

All subjects consume a weight-maintaining diet containing 200-250 g of carbohydrate/day for at least three days before studies. Body weight must be stable in all subjects for at least 1 month before studies. No subject should participate in any heavy exercise. Each subject gives informed written consent before participating in the research, which was approved by the Human Investigation Committee of the Verona City Hospital. Measurements of standard clinical phenotypes are collected in all patients. Other diabetes related phenotypes may be collected if their determination is available.

Metabolic tests are carried out on two separate days in random order. On both days, patients are admitted to the Metabolic Clinic Research Center at 07:30 after an overnight fast. All studies are carried out in a quiet, temperature controlled (22° C) room. On one day an oral glucose tolerance test (OGTT) (75 g) is performed to assess beta cell function. On a separate day, a euglycemic insulin clamp is performed to assess insulin sensitivity.

When age of onset and distribution of the disease in the pedigree suggest a potentially monogenic disorder, the relatives of the proband are asked to participate in the study by allowing the collection of standard clinical information and of a fasting blood sample for genetic and phenotypic determinations.

-OGTT: For ethical reasons, the OGTT cannot performed in patients presenting with fasting plasma glucose higher than 15 mmol/l. During the entire test patients are sitting in a comfortable cardiac chair. One teflon (21 g) venous catheter is inserted into an antecubital vein for blood sampling and kept patent with heparinized normal saline solution. After a 30' rest to establish baseline and after collecting a 20 cc blood sample for leukocyte DNA extraction, at time = 0' subjects ingest 75 g of glucose in 300 ml of water over 5 min. Blood samples to measure glucose, C-peptide and insulin concentrations are collected at times -10', 0', +15', +30', +45', +60', +90', +120', +150', +180', +210' and +240', +270' and +300'. Urines are collected to measure glycosuria.

-Euglycemic Insulin Clamp: During the entire test patients are lying in bed. One teflon catheter is introduced into an antecubital vein for the infusion of test substances. Another teflon catheter is placed retrogradely into a wrist vein for sampling arterialized venous blood, according to the "hot box" technique. After a 30' rest in bed to establish baseline, indirect calorimetry (at least 40') is performed. At the end of calorimetric measures, baseline blood samples are collected and a standard euglycemic insulin clamp is carried out. After an insulin intravenous prime of 4.8 pmol/min/m^2 BSA and a subsequent continuous infusion of 240 pmol/min/m^2 BSA, plasma glucose is allowed to decline until it reaches 5.5 mmol/l, after which glucose clamping starts with a glucose concentration goal of 5 mmol/l. The duration of the glucose clamp is at least of 120', but it is prolonged, if and as needed, to ensure at least 60' of insulin clamp at euglycemia in each patient. Timed blood samples were collected to measure hormone and substrate levels. In the last 45' of the clamp indirect calorimetry is repeated to assess substrate oxidation and energy production rates. Urine is collected to measure urea excretion rate.

In both metabolic tests, all blood samples are collected in pre-chilled tubes and readily spun at 1,500 g. Plasma and serum specimens are stored at -80° C.

-Analytical procedures: Plasma glucose concentration is measured in duplicate at bedside. Serum C-peptide and insulin concentrations are measured by chemiluminescence. Glycated hemoglobin and serum lipids were measured by standard in-house methods. GAD-antibodies are measured by immunoradiometry (CentAK, Medipan, Germany), according to manufacturer's instructions.

-Genotyping: A leukocyte DNA sample is collected in each subject and the DNA is extracted through standard salting out method. Genotyping is performed by RFLP (Restriction Fragment Length Polymorphism), which consists in a PCR (Polymerase Chain Reaction) followed by proper enzymatic digestion and resolution on agarose gel. Alternatively, it is performed were assessed by the high-throughput genotyping Veracode technique (Illumina Inc, CA), applying the GoldenGate Genotyping Assay according to manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, whose diagnosis has been made in the last six months before the first access to the Division of Endocrinology and Metabolic Diseases of University of Verona School of Medicine;
* Relatives of patients with potentially monogenic newly diagnosed type 2 diabetes

Exclusion Criteria:

* Age > 75 years
* Non-Italian ancestry
* Insulin treatment
* Presence of anti-GAD antibodies
* Malignancies
* Any condition severely impairing liver and/or kidney function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A: all patients referred to the Division of Endocrinology and Metabolic Diseases of University of Verona School of Medicine, whose diabetes has been diagnosed in the last six months, are asked to participate in this research.
  Group B: Relatives of patients with potentially monogenic newly diagnosed type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2003-10; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Genetic basis of beta cell function | Baseline and during the 75 g oral glucose challenge. Subjects will be followed for the duration of their stay in the Metabolic Clinical Research Center (average expected stay: 6 hours)
  Investigators genotype diabetes risk loci and relate them to two main beta cell metrics, after correction for insulin sensitivity:
  1. Derivative control of beta cell function: it is the amount of insulin secreted in response to a rate of glucose increase of 1 mmol/l per min which lasts for 1 minute;
  2. Proportional control of beta cell function: it is the stimulus-response curve linking glucose concentration (x-axis) to insulin secretion rate (y-axis) at the preselected glucose concentrations of 5.5, 8.0, 11.0, 15.0, and 20.0 mmol/liter.

SECONDARY OUTCOMES:
Genetic basis of insulin sensitivity | Baseline and during the euglycemic insulin clamp. Subjects will be followed for the duration of their stay in the Metabolic Clinical Research Center (average stay: 4 hours)
  Investigators genotype diabetes risk loci and relate them, after correcting for the influence of other genetic and nongenetic modifiers, to one metric of clamp derived insulin sensitivity:
  1. M value, which quantifies whole body net glucose disposal during euglycemic hyperinsulinemia

CONTACTS AND LOCATIONS:
Overall Officials: Enzo Bonora, MD PhD, Study Chair — Section of Endocrinology, Diabetes and Metabolism - Department of Medicine, University of Verona and Azienda Ospedaliera Universitaria Integrata, Verona, Italy; Riccardo C Bonadonna, MD, Principal Investigator — Section of Endocrinology, Diabetes and Metabolism - Department of Medicine, University of Verona and Azienda Ospedaliera Universitaria Integrata, Verona, Italy
Locations (1):
- Division of Endocrinology and Metabolic Diseases - University Hospital of Verona, Verona, Italy

REFERENCES:
- [Derived] Bonora E, Trombetta M, Dauriz M, Brangani C, Cacciatori V, Negri C, Pichiri I, Stoico V, Rinaldi E, Da Prato G, Boselli ML, Santi L, Moschetta F, Zardini M, Bonadonna RC. Insulin resistance and beta-cell dysfunction in newly diagnosed type 2 diabetes: Expression, aggregation and predominance. Verona Newly Diagnosed Type 2 Diabetes Study 10. Diabetes Metab Res Rev. 2022 Oct;38(7):e3558. doi: 10.1002/dmrr.3558. Epub 2022 Jul 5. PMID 35717608
- [Derived] Bonora E, Trombetta M, Dauriz M, Travia D, Cacciatori V, Brangani C, Negri C, Perrone F, Pichiri I, Stoico V, Zoppini G, Rinaldi E, Da Prato G, Boselli ML, Santi L, Moschetta F, Zardini M, Bonadonna RC. Chronic complications in patients with newly diagnosed type 2 diabetes: prevalence and related metabolic and clinical features: the Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) 9. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001549. doi: 10.1136/bmjdrc-2020-001549. PMID 32819978
- [Derived] Trombetta M, Dauriz M, Bonetti S, Travia D, Boselli L, Santi L, Bonora E, Bonadonna RC. Is common genetic variation at IRS1, ENPP1 and TRIB3 loci associated with cardiometabolic phenotypes in type 2 diabetes? An exploratory analysis of the Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) 5. Nutr Metab Cardiovasc Dis. 2016 Mar;26(3):232-8. doi: 10.1016/j.numecd.2016.01.002. Epub 2016 Jan 14. PMID 26868433
- [Derived] Dauriz M, Trombetta M, Boselli L, Santi L, Brangani C, Pichiri I, Bonora E, Bonadonna RC. Interleukin-6 as a potential positive modulator of human beta-cell function: an exploratory analysis-the Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) 6. Acta Diabetol. 2016 Jun;53(3):393-402. doi: 10.1007/s00592-015-0807-z. Epub 2015 Nov 4. PMID 26538364
- [Derived] Zoppini G, Cacciatori V, Raimondo D, Gemma M, Trombetta M, Dauriz M, Brangani C, Pichiri I, Negri C, Stoico V, Bergamini C, Targher G, Santi L, Thomaseth K, Bellavere F, Bonadonna RC, Bonora E. Prevalence of Cardiovascular Autonomic Neuropathy in a Cohort of Patients With Newly Diagnosed Type 2 Diabetes: The Verona Newly Diagnosed Type 2 Diabetes Study (VNDS). Diabetes Care. 2015 Aug;38(8):1487-93. doi: 10.2337/dc15-0081. Epub 2015 Jun 11. PMID 26068862